CLINICAL TRIAL: NCT03163004
Title: Implementing Standing Desks in Primary and Secondary Schools to Reduce Sedentary Time: Effect and Process Evaluation.
Brief Title: Implementation of Standing Desks at School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Principal Investigator, Vakgroepsport, Prof. Dr. Greet Cardon, University Ghent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWO13/PDO/191 second term
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Health Behavior
Keywords: Sedentary behavior
MeSH Terms: conditions — Health Behavior; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: One intervention and one control condition
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Implementation of standing desks in the classroom
  Interventions: Behavioral: Implementation of standing desks
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Implementation of standing desks — Three standing desks will be introduced to the classroom
  Arms: Intervention group

SUMMARY:
Since sedentary time is related to various health outcomes and is already highly prevalent in childhood and adolescence, effective strategies are needed to tackle this health problem. Children and adolescents spend the majority of the day in a classroom while sitting at a desk. Therefore, the classroom is an important setting for implementing specific strategies to reduce sedentary time.

One of the strategies that gained more attention during the past years is replacing traditional desks and chairs with standing desks.

This project evaluates the implementation of standing desks in primary and secondary schools via a clustered randomized controlled trial using an intervention and control condition. Effects on sedentary time during in class, sedentary activities during leisure time, breaks in sedentary time, and related determinants (secondary outcomes) are evaluated.

Next to effect evaluation, it is also equally important to evaluate how teachers and pupils perceive this change in the classroom environment. Both groups need to be positive in order to obtain the adoption and sustainability. Therefore, focus groups with pupils and interviews with teachers are conducted, with a specific focus on the perceived barriers. Moreover, the process evaluation is conducted quantitatively as well by using questionnaires in pupils and teachers.

The project results will lead to recommendations on how to broadly implement standing desks into primary and secondary schools.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pupils of primary schools (5th grade) and secondary schools (10th grade)

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 343 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Decrease in children's sedentary time during school hours | One schoolyear
  In the questionnaire, following item was used to subjectively assess the outcome: 'On average how many hours do you spent sedentary in class?' Answer categories ranged from 'None' to 'More than 7 hours per day'. In addition, a subsample wore an ActivPAL inclinometer to objectively measure sedentary time. This thigh-worn device uses accelerometer-derived information about thigh position to calculate the outcome.

SECONDARY OUTCOMES:
Possible decrease in TV time on week- and weekend days | One schoolyear
  In the questionnaire, children and adolescents were asked on average how many hours they spent in front of a television, separately for week- and weekend days. Answer categories ranged from 'Non' to 'More than 4 hours per day'. The items are derived from the reliable and valid ENERGY-questionnaire.
Possible decrease in computer time on week- and weekend days | One schoolyear
  In the questionnaire, children and adolescents were asked on average how many hours they spent in front of a computer, separately for week- and weekend days. Answer categories ranged from 'Non' to 'More than 4 hours per day'. The items are derived from the reliable and valid ENERGY-questionnaire.
Increase in the number of breaks in sedentary activities | One schoolyear
  In the questionnaire, children and adolescents were asked on average, how many times they interrupt their TV time, computer time and sitting during school hours. Answer categories ranged from '0' to '4 times or more per hour'. The items were derived from the ENERGY-questionnaire.
Improvement of determinants related to breaking up sedentary activities | One schoolyear
  In the questionnaire, questions were added on attitude, self-efficacy, preferences and habits related to breaking up sedentary activities, with answer categories ranging from 'Totally agree' to 'Totally disagree'. The items were derived from the ENERGY-questionnaire
Improvement in school well-being | One schoolyear
  Three school-related variables (i.e. relationship with classmates, involvement in organising school activities, and relationship with teachers) were assessed in the questionnaire using items from the Flemish Health Behaviour in School-Aged Children questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Department of Movement and Sports Sciences, Ghent, Belgium

REFERENCES:
- [Derived] Neil-Sztramko SE, Caldwell H, Dobbins M. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6 to 18. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD007651. doi: 10.1002/14651858.CD007651.pub3. PMID 34555181
- [Derived] Verloigne M, Ridgers ND, De Bourdeaudhuij I, Cardon G. Effect and process evaluation of implementing standing desks in primary and secondary schools in Belgium: a cluster-randomised controlled trial. Int J Behav Nutr Phys Act. 2018 Sep 27;15(1):94. doi: 10.1186/s12966-018-0726-9. PMID 30261883